CLINICAL TRIAL: NCT03378232
Title: EPA and DHA Regulation of Blood Triglycerides, Resting Metabolic Rate and Blood Markers of Cardiometabolic Health.
Brief Title: Cardiometabolic Benefits of Omega-3 Polyunsaturated Fatty Acids
Acronym: TGIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government)
Responsible Party: Principal Investigator, David M Mutch, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The Goodness In Fish Oil
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Disease
Keywords: DHA; EPA; fatty acids; blood pressure; resting metabolic rate; blood lipids; muscle sympathetic nerve activity (MSNA)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant as well as student investigators were blinded to the treatment randomization.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Olive Oil (Placebo Comparator): Placebo supplement with olive oil
  Interventions: Dietary Supplement: Placebo Olive Oil
- High EPA Supplement (Experimental): Supplements providing up to 3g per day of Omega-3, with increased EPA
  Interventions: Dietary Supplement: High EPA Supplement
- High DHA Supplement (Experimental): Supplements providing up to 3g per day of Omega-3, with increased DHA
  Interventions: Dietary Supplement: High DHA Supplement

INTERVENTIONS:
Dietary Supplement: Placebo Olive Oil — Each participant was instructed to consume the dietary supplement on a daily basis for 12 weeks.
  Arms: Placebo Olive Oil
Dietary Supplement: High EPA Supplement — Each participant was instructed to consume assigned dietary supplement on a daily basis for 12 weeks.
  Arms: High EPA Supplement
Dietary Supplement: High DHA Supplement — Each participant was instructed to consume assigned dietary supplement on a daily basis for 12 weeks.
  Arms: High DHA Supplement

SUMMARY:
Omega 3 fatty acids have been shown to provide a number of cardiometabolic benefits in both healthy and at risk populations. Specifically, the daily consumption of fish oil supplements has been reported to reduce blood triglyceride levels, and influence glucose homeostasis and whole-body inflammation. Furthermore, a number of cardiovascular effects (i.e. reduced blood pressure, reduced coagulation) have been found to result from omega-3 consumption, as well as influencing energy expenditure (i.e. resting metabolic rate). The goal of this study is to examine the cardiometabolic and cardiovascular effects that result from long-term consumption of omega-3 fatty acids.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and type 2 diabetes (T2D) are major contributors to healthcare costs in Canada. A cluster of cardiometabolic risk factors including insulin resistance, dyslipidemia, hypertension, and abdominal obesity increases the risk of developing the aforementioned diseases. While drugs can help to treat or slow the development of cardiometabolic problems, they are not always effective and in some instances can have adverse effects on a patient's health. In comparison, changing, modifying or improving dietary habits is now recognized as a safe and effective way to help reduce the risk of developing CVD, as well as treat CVD and T2D. The consumption of omega-3 fatty acids (FAs) is highly recommended due to their known benefits for health and development; however, considerable variability exists in the literature regarding the benefits of omega-3 FAs. This variability stems from differences in study design; differing in dosage, duration of supplementation, population studied, sample size, as well as the amounts of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) used in supplements. The current study will investigate the effects of EPA and DHA on markers of cardiometabolic and cardiovascular health in young adults.

To assess the effectiveness of EPA and DHA on markers of cardiometabolic health, including

1. blood lipids, such as triglycerides, total cholesterol, high-density lipoprotein (HDL) and low-density lipoprotein (LDL) levels
2. markers of inflammation, such as high-sensitivity C-reactive protein (hs-CRP) and other circulating cytokines
3. whole-body glucose and insulin levels
4. resting metabolic rate
5. blood pressure and muscle sympathetic nerve activity

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years
* Healthy

Exclusion Criteria:

* Younger than 18 years
* Older than 30 years
* Allergic to fish and/or shellfish or gelatin
* High consumption of omega-3 fats (either fatty fish or dietary supplements)
* Chronic or communicable diseases
* Anticipated change in lifestyle (moving to a new house, starting a new fitness routine).
* Discomfort giving blood
* Use of lipid-controlling medication, including cholesterol lowering drugs (statins), fatty acid/triglyceride altering (fibrates) or any other drug known to have lipid altering effects, such as ezetimibe, colesevelam, torcetrapib, avasimibe, and implitapide
* Chronic use of anti-inflammatory medications
* Pregnant, or is planning to become pregnant during the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Omega-3 Index | CHANGE from Baseline at 12 weeks
  Omega-3 Index, as determined by measuring omega-3 fats in red blood cells using gas chromatography

SECONDARY OUTCOMES:
Triglycerides | CHANGE from Baseline at 12 weeks
  Fasted serum triglycerides (mmol/L)
High-sensitivity C-Reactive Protein (hs-CRP) | CHANGE from Baseline at 12 weeks
  Blood hs-CRP levels
Energy Expenditure | CHANGE from Baseline at 12 weeks
  Resting Metabolic Rate
Blood Pressure | CHANGE from Baseline at 12 weeks
  Both systolic and diastolic blood pressure will be assessed
Muscle sympathetic nerve activity (MSNA) | Change from Baseline at 12 weeks
  Fibular nerve microneurography

CONTACTS AND LOCATIONS:
Overall Officials: David M Mutch, PhD, Principal Investigator — University of Guelph; Phillip Millar, PhD, Principal Investigator — University of Guelph; Lawrence Spriet, PhD, Principal Investigator — University of Guelph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roke K, Mutch DM. The role of FADS1/2 polymorphisms on cardiometabolic markers and fatty acid profiles in young adults consuming fish oil supplements. Nutrients. 2014 Jun 16;6(6):2290-304. doi: 10.3390/nu6062290. PMID 24936800
- [Background] Roke K, Jannas-Vela S, Spriet LL, Mutch DM. FADS2 genotype influences whole-body resting fat oxidation in young adult men. Appl Physiol Nutr Metab. 2016 Jul;41(7):791-4. doi: 10.1139/apnm-2016-0043. Epub 2016 Mar 16. PMID 27144909
- [Background] Miller PE, Van Elswyk M, Alexander DD. Long-chain omega-3 fatty acids eicosapentaenoic acid and docosahexaenoic acid and blood pressure: a meta-analysis of randomized controlled trials. Am J Hypertens. 2014 Jul;27(7):885-96. doi: 10.1093/ajh/hpu024. Epub 2014 Mar 6. PMID 24610882
- [Background] Merino DM, Ma DW, Mutch DM. Genetic variation in lipid desaturases and its impact on the development of human disease. Lipids Health Dis. 2010 Jun 18;9:63. doi: 10.1186/1476-511X-9-63. PMID 20565855
- [Background] Klingel SL, Roke K, Hidalgo B, Aslibekyan S, Straka RJ, An P, Province MA, Hopkins PN, Arnett DK, Ordovas JM, Lai CQ, Mutch DM. Sex Differences in Blood HDL-c, the Total Cholesterol/HDL-c Ratio, and Palmitoleic Acid are Not Associated with Variants in Common Candidate Genes. Lipids. 2017 Dec;52(12):969-980. doi: 10.1007/s11745-017-4307-5. Epub 2017 Oct 27. PMID 29080057
- [Derived] Metherel AH, Valenzuela R, Klievik BJ, Cisbani G, Rotarescu RD, Gonzalez-Soto M, Cruciani-Guglielmacci C, Laye S, Magnan C, Mutch DM, Bazinet RP. Dietary docosahexaenoic acid (DHA) downregulates liver DHA synthesis by inhibiting eicosapentaenoic acid elongation. J Lipid Res. 2024 Jun;65(6):100548. doi: 10.1016/j.jlr.2024.100548. Epub 2024 Apr 20. PMID 38649096
- [Derived] Klingel SL, Metherel AH, Irfan M, Rajna A, Chabowski A, Bazinet RP, Mutch DM. EPA and DHA have divergent effects on serum triglycerides and lipogenesis, but similar effects on lipoprotein lipase activity: a randomized controlled trial. Am J Clin Nutr. 2019 Dec 1;110(6):1502-1509. doi: 10.1093/ajcn/nqz234. PMID 31535138
- [Derived] Metherel AH, Irfan M, Klingel SL, Mutch DM, Bazinet RP. Compound-specific isotope analysis reveals no retroconversion of DHA to EPA but substantial conversion of EPA to DHA following supplementation: a randomized control trial. Am J Clin Nutr. 2019 Oct 1;110(4):823-831. doi: 10.1093/ajcn/nqz097. PMID 31204771